CLINICAL TRIAL: NCT01914731
Title: Fecal Microbiota Transplant (FMT) for Relapsing Clostridium Difficile Infection in Adults and Children Using a Frozen Encapsulated Inoculum
Brief Title: Fecal Microbiota Transplant for Relapsing Clostridium Difficile Infection in Adults and Children Using a Frozen Encapsulated Inoculum
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-P-001355
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Clostridium Difficile Infection
Keywords: Fecal Microbiota Transplant; Clostridium difficile; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capsule (Experimental): Fecal microbiota transplant ("stool transplant") from healthy, unrelated donor via frozen capsule
  Interventions: Drug: Fecal Microbiota Transplant

INTERVENTIONS:
Drug: Fecal Microbiota Transplant — Reconstitution of normal flora by a "stool transplant" from a healthy individual to a C. difficile - infected recipient via frozen capsule
  Other Names: Poop transplant; Fecal bacteriotherapy

SUMMARY:
Fecal microbiota transplantation (FMT) is the reconstitution of normal flora by a "stool transplant" from a healthy individual to a C. difficile-infected recipient, and has long been a successful approach to recurrent/refractory C. difficile. The purpose of this project is to generate a frozen FMT inoculum from well-screened healthy volunteer donors which can be used repeatedly, particularly in those who do not have a healthy intimate partner or other related donor. Delivery of FMT has been performed colonoscopically, by fecal retention enema, or by the nasogastric route. This study will evaluate the safety and secondarily the efficacy of an inoculum administered by frozen orally-administered capsules.

Subjects with recurrent/relapsing C. difficile infection will receive FMT via oral capsules

The primary endpoint is assessment of safety as measured by clinical events (GI, procedural, systemic). Efficacy will be defined as a resolution of diarrhea off antibiotics for C. difficile, in the absence of a need for OTHER systemic antibiotics, i.e. resumption of a normal bowel status for the individual. Secondary efficacy endpoints include weight, subjective well-being and relative clinical improvement per standardized questionnaire, and subject qualitative assessment of, and satisfaction with, the transplant procedures. Subjects will be monitored for clinical safety by history and standard exams and the follow-up questionnaire as well as followed closely by phone and in person.

ELIGIBILITY:
Inclusion criteria

* Patients with refractory, recurrent or relapsing C. difficile infection (CDI) defined as EITHER:

  * At least three episodes of mild-to-moderate CDI
  * At least two episodes of severe CDI resulting in hospitalization and associated with significant morbidity
  * One protracted episode of CDI, defined as at least 3 weeks of ongoing Grade 3 severe symptoms of CDI despite standard antimicrobial therapy for CDI
  * We expect that most, but not all, subjects will have tried and failed a taper of vancomycin.
* Willingness to accept risk of unrelated donor stool
* Age 7 and above. Seven is chosen as a lower limit based upon the legal age of assent. Based on the literature, most children aged 7 and above can be taught to swallow even large capsules through simple coaching techniques
* Able to consent for self, or parental assent/child assent as age appropriate

Exclusion criteria

* Delayed gastric emptying syndrome
* Known chronic aspiration
* Swallowing dysfunction or oral-motor dyscoordination.
* Inability or unwillingness to swallow multiple large capsules
* Pregnant women
* Patients with an acute illness unrelated to CDI or an acute exacerbation of underlying comorbid condition
* Patients with comorbidities associated with increased risk of serious infection following bacterial translocation, including but not limited to:

  * subjects on major immunosuppressive agents including high dose corticosteroids, calcineurin inhibitors, mTOR inhibitors, lymphocyte depleting biologic agents, anti-TNF agents, and others; chemotherapeutic anti-neoplastic agents*
  * Patients with decompensated liver cirrhosis, advanced HIV/AIDS, recent bone marrow transplant, hypoglobulinemia or other cause of severe immunodeficiency*
* Patients with a history of significant allergy to foods not excluded from the donor diet

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 6 months post-FMT
  Safety is assessed by clinical symptoms, exam, signs (GI and systemic)

SECONDARY OUTCOMES:
Efficacy | Up to 2 months post-FMT
  Efficacy is defined as resolution of C. Difficile signs and symptoms off antibiotics for C. difficile

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hohmann, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- See also: JAMA paper — http://www.ncbi.nlm.nih.gov/pubmed?term=JAMA%5BJour%5D+AND+hohmann%5Bauthor%5D&cmd=detailssearch